CLINICAL TRIAL: NCT07350135
Title: Impact of Sodium Supplementation on Postnatal Growth of Premature Neonates: a Randomised Controlled Clinical Trial
Brief Title: Sodium Supplementation and Growth in Premature Neonates
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MD122a/2025
Record Dates: First submitted 2025-11-20; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Sodium Supplementation and Growth in Premature Neonates
MeSH Terms: interventions — Urination

STUDY DESIGN:
Intervention Model Description: at least 74 premature neonates (37 in each group) By using Power Analysis and Sample Size Software (PASS 15) (Version 15.0.10) for sample size calculation, setting power at 80%, significance level 0.05 and after reviewing previous study results [9] showing that among preterm infants, infants who received sodium supplementation had greater Percentage increase from birth at 6 weeks of age than those who do not (194.9 + 18 versus 182.6 + 19 respectively); Based on that, a sample size of at least 74 Preterm infants (gestational age <34 weeks and birth weight <2500 gm) randomly assigned according to gender and gestational age into 2 groups (37 neonate in each group) will be needed.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): - Group A: will receive sodium supplementation with a moderate dose (4 mEq/kg/day) above basic maintenance requirements starting from 7 days to 28 days after birth.
  Interventions: Drug: Sodium supplementation guided by serum sodium and fraction sodium in urine
- - Group B: control group (No Intervention): - Group B: control group will not receive above basic maintenance requirements

INTERVENTIONS:
Drug: Sodium supplementation guided by serum sodium and fraction sodium in urine — The Study population will be stratified according to gender and gestational age and randomly assigned into 2 groups:
  * Group A: will receive sodium supplementation with a moderate dose (4 mEq/kg/day) above basic maintenance requirements starting from 7 days to 28 days after birth. Sodium will be supplemented in the form of hypertonic saline provided either parenteral (added to maintenance intravenous fluid) or enteral, if oral intake exceeds 100 ml/kg/day (divided and added to feds every 6 hours) [9] (withhold supplementation if the serum sodium reaches 150 mmol/L, or development of vomiting or diarrhea with oral supplementation).
  * Group B: control group will receive basic maintenance requirements of the sodium supplementation (3mEq/kg/day).
  Arms: Group A

SUMMARY:
Primary aim: to assess the impact of late (≥7 days postnatal) sodium supplementation of premature neonates with birth weight less than 2500 gm on their postnatal short-term catch-up growth.

Secondary aim: to find out the effect of this sodium supplementation on fractional excretion of sodium, hemodynamics and prematurity-related short-term neonatal outcomes including morbidities and morality.

DETAILED DESCRIPTION:
Preterm birth is a global health problem and the primary contributor to neonatal mortality and morbidity [2].

Poor growth after preterm birth is challenging and arises from a combination of various factors, including nutritional needs, hormonal abnormalities, central nervous system damage, feeding difficulties, and administration of drugs that affect nutrient metabolism [3].

Typically, weight gain in the neonatal period begins after the first week of life, considered a period of physiological weight loss. With a mean period of 10.6 days, preterm neonates experience an average weight gain of 16.7 g/kg per day after reaching their birth weight [4].

The shift from the intra- to the extrauterine environment is associated with significant alternations in water and electrolytes, especially sodium homeostasis. In the early phase, this is primarily marked by decreased extracellular fluid volume and sodium loss. This adaptation becomes considerably more complex in premature infants due to immature kidneys, which lack full regulatory functionality and increased transdermal water loss [5]. Consequently, premature infants are at risk to hypernatremia early in life. In contrast, after the initial postnatal period with skin maturation, these infants become susceptible to hyponatremia because of the inability of the premature kidney to retain salt [6]. This often necessitates high sodium substitution to ensure adequate growth [5].

Sodium plays a crucial role for protein synthesis, bone mineralization, maintenance of extracellular space, and enabling the transport of glucose across the cell membranes [7]. Sodium can be considered a growth factor that stimulates protein synthesis and increase cell mass, and thus inadequate sodium intake can lead to chronic sodium depletion and thus growth failure [1].

The European Society of Pediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN) Committee of Nutrition recently issued updated recommendations for sodium intake of 3-8 mEq/kg/day for preterm infants during the first few months of birth[1,8].

ELIGIBILITY:
Inclusion Criteria:

* Preterm from 28 to 34 weeks gestation, admitted to NICU.
* Birth weight (<2500 gm). Postnatal age ≥7 days

Exclusion Criteria:

* - Major congenital malformations.
* Congenital heart disease
* Renal insufficiency (defined as an increase in serum creatinine by ≥0.5 mg/dL/d, urine output <0.5 mL/kg/h) [10].
* Disease states characterized by fluid retention: as cardiac, hepatic or renal.
* Receiving diuretic therapy.
* Full term less than 2500 gm.

Ages: 7 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2025-11-06 (Actual); Primary Completion 2028-11-06 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
follow up weight of preterm for 6 weeks | since birth till the age of 6 weeks postnatally.
  measuring birth weight of the neonate Initially and then twice weekly in grams (g) and z-scores will be calculated using the Fenton Preterm Growth Chart for boys or girls. This will continue till the age of 6 weeks postnatal life.

SECONDARY OUTCOMES:
Laboratory studies | twice weekly till 6 weeks post natal
  1. Serum sodium concentration: initial level, then twice weekly to report hyponatremia (defined as serum sodium <130 mmol/L) or hypernatremia (defined as serum sodium ≥ 150 mmol/L).
  2. Fractional Excretion of Sodium: initial level, then after two weeks from sodium supplementation calculated by measuring creatinine and sodium levels in the blood and urine simultaneously [(urinary sodium × serum creatinine)/ (urinary creatinine × serum sodium)×100).

CONTACTS AND LOCATIONS:
Locations (1):
- Eldemerdash Hospital, Cairo, Egypt